CLINICAL TRIAL: NCT03659825
Title: Ketone Esters for Optimization of Cognitive Performance in Hypoxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HVMN Inc (Industry)
Collaborators: Florida Institute for Human and Machine Cognition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KEHYPOX18
Record Dates: First submitted 2018-08-14; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Hypoxia; Ketosis
MeSH Terms: conditions — Hypoxia; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Intervention Model Description: Young healthy adults.
Who Masked: Participant, Investigator
Masking Description: Study drinks will be matched for taste and appearance. Investigator preparing and administering the drink will not carry out the testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo + Normoxia (Placebo Comparator): Taste, volume and appearance matched drink given before cognitive testing in normoxia
  Interventions: Dietary Supplement: Taste Matched Placebo
- Placebo + Hypoxia (Placebo Comparator): Taste, volume and appearance matched drink given before cognitive testing in hypoxia
  Interventions: Dietary Supplement: Taste Matched Placebo; Other: Hypoxic exposure
- Ketone Ester + Normoxia (Experimental): Ketone ester drink given before cognitive testing in normoxia
  Interventions: Dietary Supplement: Ketone Ester
- Ketone Ester + Hypoxia (Experimental): Ketone ester drink given before cognitive testing in hypoxia
  Interventions: Dietary Supplement: Ketone Ester; Other: Hypoxic exposure

INTERVENTIONS:
Dietary Supplement: Ketone Ester — Flavored sports drink containing deltaG (betahydroxybutyrate monoester) as the sole active ingredient, diluted with water.
  Other Names: HVMN Ketone
  Arms: Ketone Ester + Hypoxia; Ketone Ester + Normoxia
Dietary Supplement: Taste Matched Placebo — Placebo that tastes similar to active intervention
  Arms: Placebo + Hypoxia; Placebo + Normoxia
Other: Hypoxic exposure — Participants will breath through a mask to provide the amount of oxygen typically seen at 16-17,000ft of altitude.
  Arms: Ketone Ester + Hypoxia; Placebo + Hypoxia

SUMMARY:
This study will investigate the effects of ketone ester drinks on cognitive performance in hypoxia.

DETAILED DESCRIPTION:
In the setting of altitude-induced hypoxia, cognitive capacity degrades and can compromise both individual and team performance. This degradation is linked to falling brain energy (ATP) levels and an increased reliance on anaerobic energy production from glucose. Ketone bodies are the evolutionary alternative substrate to glucose for brain metabolic requirements; previous studies have shown that the presence of elevated ketone bodies (ketosis) maintains brain ATP levels and reduce cerebral anaerobic glycolysis during hypoxia. Ketosis can be achieved when fasting or following a ketogenic diet; however, these approaches are impractical. Exogenous ketone ester supplementation allows for rapid (< 30 mins) and significant elevation of blood ketone levels without the need to maintain a diet or fast.

HVMN, in collaboration with researchers at IHMC, proposes a study to investigate the effects of consuming an FDA-approved ketone ester 'food' on cognitive performance in the setting of hypoxia. For the proposed 4-arm within-subject study, participants will complete a cognitive performance test battery under the conditions of normoxia and then hypoxia following consumption of a ketone ester drink or a placebo drink (N.B for each study drink cognitive performance in both hypoxia and normoxia will be assessed in ONE visit):

VISIT A:

Arm1: Normoxia + Placebo Arm 2: Hypoxia + Placebo

VISIT B:

Arm 3: Normoxia + Ketone ester Arm 4: Hypoxia + Ketone ester

The investigators hypothesize that ketone ester supplementation will attenuate hypoxia-induced deterioration of operator cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Pass medical examination on enrollment.

Exclusion Criteria:

* Active smoker, substance abuse.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Performance- Visual Acuity | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (visual acuity) will be assessed using the RightEye testing system (https://www.righteye.com).
Change in Cognitive Performance- Contrast Sensitivity | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (contrast sensitivity) will be assessed using the RightEye testing system (https://www.righteye.com).
Change in Cognitive Performance- Choice Reaction Time | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (choice reaction time) will be assessed using both the RightEye testing system (https://www.righteye.com) and the DANA testing system (http://www.danabrainvital.com).
Change in Cognitive Performance- Eye Tracking- Smooth Pursuit | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (eye tracking) will be assessed by looking for smooth pursuit (horizontal and vertical) using the RightEye testing system (https://www.righteye.com).
Change in Cognitive Performance- Eye Tracking- Saccades | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (eye tracking) will be assessed by looking at saccade speed (horizontal and vertical) using the RightEye testing system (https://www.righteye.com).
Change in Cognitive Performance- Simple Reaction Time | Measured 3 times (baseline [time = 0 min], during normoxia [time = 30-60 min post study drink 1] and during hypoxia [30-60 min post study drink 2]) in each of the two test visits.
  Cognitive performance (simple reaction time) will be assessed using both the RightEye testing system (https://www.righteye.com) and the DANA testing system (http://www.danabrainvital.com).

SECONDARY OUTCOMES:
Change in Grip Strength | Measured 3 times (baseline [time = 0 min], after normoxia [60 min post study drink 1] and after hypoxia [60 min post study drink 2]) in each of the two test visits.
  Grip strength will be measured using a
Change in blood ketone levels | Measured 5 times at regular intervals through each of the two study visits. [time (min) = 0, 30, 75, 105, 150]
  Blood ketone levels will be measured in a finger prick blood samples using a clinical grade, handheld glucose/ketone meter (Abott Diabetes Care).
Change in blood glucose levels | Measured 5 times at regular intervals through each of the two study visits. [time (min) = 0, 30, 75, 105, 150]
  Blood glucose levels will be measured in a finger prick blood samples using a clinical grade, handheld glucose/ketone meter (Abott Diabetes Care).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Suzuki M, Suzuki M, Sato K, Dohi S, Sato T, Matsuura A, Hiraide A. Effect of beta-hydroxybutyrate, a cerebral function improving agent, on cerebral hypoxia, anoxia and ischemia in mice and rats. Jpn J Pharmacol. 2001 Oct;87(2):143-50. doi: 10.1254/jjp.87.143. PMID 11700013
- [Background] Kirsch JR, D'Alecy LG, Mongroo PB. Butanediol induced ketosis increases tolerance to hypoxia in the mouse. Stroke. 1980 Sep-Oct;11(5):506-13. doi: 10.1161/01.str.11.5.506. PMID 6775394
- [Background] Xu K, Sun X, Eroku BO, Tsipis CP, Puchowicz MA, LaManna JC. Diet-induced ketosis improves cognitive performance in aged rats. Adv Exp Med Biol. 2010;662:71-5. doi: 10.1007/978-1-4419-1241-1_9. PMID 20204773
- See also: HVMN product website — https://hvmn.com